CLINICAL TRIAL: NCT02943967
Title: Two Years Follow up of Corneal Cor Cross-linking and Refractive Surface Ablation in Patients With Asymmetric Corneal Topography
Brief Title: Corneal Cross-linking and Refractive Surface Ablation in Patients With Asymmetric Corneas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Mauro Campos, medical doctor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2088/88
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Surgical Procedure, Unspecified
Keywords: Refractive Surgical Procedures; Photorefractive Keratectomy; Aberrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CXL + PRK group (Active Comparator): Corneal cross-linking surgery is perfomed in one eye : deepithelization of the cornea and instillation of 0,1% riboflavin (ophthalmos - Brazil) for 30 minutes and UVA for irradiated for 30 minutes with ultraviolet-A of 365nm light with an irradiance of 3 mW/cm2 using Xlink (Opto - São Carlos) Photorefractive keratotomy will be perfomed in the same eye using excimer laser Ladarvision (Alcon - USA) with 0,02 % mitomicin for 30 seconds (Ophthalmos - Brasil) simultaneously with the other eye.
  Both procedures will have the same post operative treatment :
  gatifloxacin 0,3% 6/6h for 10 days prednisolone acetate 0,12% 6/6h por 14 days
  Interventions: Procedure: CXL + PRK group
- PRK group (Active Comparator): Photorefractive keratotomy will be perfomed in the fellow eye using excimer laser Ladarvision (Alcon - USA) with 0,02 % mitomicin for 30 seconds (Ophthalmos - Brasil) simultaneously with the other eye.
  Both procedures will have the same post operative treatment :
  gatifloxacin 0,3% 6/6h for 10 days prednisolone acetate 0,12% 6/6h por 14 days
  Interventions: Procedure: PRK group

INTERVENTIONS:
Procedure: CXL + PRK group — Corneal cross-linking with subsequent photorefractive keratotomy after 6 months was performed in one eye
  Arms: CXL + PRK group
Procedure: PRK group — Photorefractive keratotomy alone was performed in contra lateral eyes
  Arms: PRK group

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of corneal cross-linking and photorefractive keratectomy for refractive correction in patients with bilateral asymmetric topography.

DETAILED DESCRIPTION:
Corneal cross-linking (CXL) by the photosensitizer, riboflavin (vitamin B2), and ultraviolet A (UVA) light increases corneal rigidity and has been described as an effective method for stabilizing the cornea in patients with progressive keratoconus. The photochemical reaction in this procedure causes the collagen to form additional covalent connections between its fibers, which stabilizes the stromal collagen fibers, improving the collagen's structure and the cornea rigidity. It is a relatively safe procedure with low rates of complications Photorefractive keratectomy (PRK) it is a traditional technique for refractive surgery. In cases of irregular corneas or re-operation normally the favorite ablation profile chosen is the guided surgery, topography guided or wavefront guided, showing better results. This technique is also relatively safe procedure with low rates of complications. One of the most unwanted complications of this surgery and also rare is corneal ectasia.

Combining PRK and CXL is already done in patients with keratoconus and suspected keratoconus.

This combined procedure uses the principle that CXL stiffen the cornea making it possible to reduce corneal thickness with PRK without weakening corneal strength. Literature show better results, in keratoconus, with simultaneous procedures. Guedj et al performed PRK in keratoconus suspects and within 5 years he did not found any corneal ectasia.

ELIGIBILITY:
Inclusion Criteria:

* bilateral asymmetric topography with inferior steepening
* corneal thickness of 440 micra at the thinnest point
* inferior-to-superior index (I-S) between 1.0D and 1.4D
* maximum keratometric steepness < 47.00D
* stable refraction more than 1 year.

Exclusion Criteria:

* forme fruste keratoconus and keratoconus
* previous eye surgery
* previous eye trauma
* confirmed pregnancy

Ages: 23 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Refractive results - spherical equivalent in diopters | 30 months

SECONDARY OUTCOMES:
Biomicroscopy findings with the slit lamp | 30 months
Visual acuity in logMar | 30 months
Aberrometric Results in root mean square | 18 months
  Only coma and spherical aberration
Topographic results in diopters | 30 months
  we will measure the increase in diopters with time
Pachymetric results in micra | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Campos, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Cheema AS, Mozayan A, Channa P. Corneal collagen crosslinking in refractive surgery. Curr Opin Ophthalmol. 2012 Jul;23(4):251-6. doi: 10.1097/ICU.0b013e3283543cbd. PMID 22569468
- [Background] Raiskup F, Theuring A, Pillunat LE, Spoerl E. Corneal collagen crosslinking with riboflavin and ultraviolet-A light in progressive keratoconus: ten-year results. J Cataract Refract Surg. 2015 Jan;41(1):41-6. doi: 10.1016/j.jcrs.2014.09.033. PMID 25532633
- [Background] Carones F, Vigo L, Scandola E, Vacchini L. Evaluation of the prophylactic use of mitomycin-C to inhibit haze formation after photorefractive keratectomy. J Cataract Refract Surg. 2002 Dec;28(12):2088-95. doi: 10.1016/s0886-3350(02)01701-7. PMID 12498842
- [Background] Randleman JB, Woodward M, Lynn MJ, Stulting RD. Risk assessment for ectasia after corneal refractive surgery. Ophthalmology. 2008 Jan;115(1):37-50. doi: 10.1016/j.ophtha.2007.03.073. Epub 2007 Jul 12. PMID 17624434
- [Background] Navas A, Ariza E, Haber A, Fermon S, Velazquez R, Suarez R. Bilateral keratectasia after photorefractive keratectomy. J Refract Surg. 2007 Nov;23(9):941-3. doi: 10.3928/1081-597X-20071101-14. PMID 18041251
- [Background] Guedj M, Saad A, Audureau E, Gatinel D. Photorefractive keratectomy in patients with suspected keratoconus: five-year follow-up. J Cataract Refract Surg. 2013 Jan;39(1):66-73. doi: 10.1016/j.jcrs.2012.08.058. Epub 2012 Oct 24. PMID 23102727
- [Background] Koller T, Mrochen M, Seiler T. Complication and failure rates after corneal crosslinking. J Cataract Refract Surg. 2009 Aug;35(8):1358-62. doi: 10.1016/j.jcrs.2009.03.035. PMID 19631120
- [Background] Abib FC, Holzchuh R, Schaefer A, Schaefer T, Godois R. The endothelial sample size analysis in corneal specular microscopy clinical examinations. Cornea. 2012 May;31(5):546-50. doi: 10.1097/ICO.0b013e3181cc7961. PMID 22333658
- [Background] Kontadakis GA, Kankariya VP, Tsoulnaras K, Pallikaris AI, Plaka A, Kymionis GD. Long-Term Comparison of Simultaneous Topography-Guided Photorefractive Keratectomy Followed by Corneal Cross-linking versus Corneal Cross-linking Alone. Ophthalmology. 2016 May;123(5):974-83. doi: 10.1016/j.ophtha.2016.01.010. Epub 2016 Feb 17. PMID 26896122
- [Background] Camellin M, Guidotti JM, Arba Mosquera S. Corneal-Wavefront guided transepithelial photorefractive keratectomy after corneal collagen cross linking in keratoconus. J Optom. 2017 Jan-Mar;10(1):52-62. doi: 10.1016/j.optom.2016.02.001. Epub 2016 Mar 21. PMID 27012841
- [Background] Shaheen MS, Shalaby Bardan A, Pinero DP, Ezzeldin H, El-Kateb M, Helaly H, Khalifa MA. Wave Front-Guided Photorefractive Keratectomy Using a High-Resolution Aberrometer After Corneal Collagen Cross-Linking in Keratoconus. Cornea. 2016 Jul;35(7):946-53. doi: 10.1097/ICO.0000000000000888. PMID 27191671
- [Background] Tomita M, Yoshida Y, Yamamoto Y, Mita M, Waring G 4th. In vivo confocal laser microscopy of morphologic changes after simultaneous LASIK and accelerated collagen crosslinking for myopia: one-year results. J Cataract Refract Surg. 2014 Jun;40(6):981-90. doi: 10.1016/j.jcrs.2013.10.044. PMID 24857441
- [Background] Guell JL, Verdaguer P, Elies D, Gris O, Manero F. Persistent stromal scar after PRK and CXL: different preoperative findings, similar complication. J Refract Surg. 2015 Mar;31(3):211-2. No abstract available. PMID 25870865